CLINICAL TRIAL: NCT07003386
Title: Exploration of the Efficacy and Mechanism of Galantamine (an Extract From Lycoris Aurea) in Treating Ischemic Stroke Based on the Neurovascular Unit
Brief Title: Exploration of the Efficacy and Mechanism of Galantamine (an Extract From Lycoris Aurea) in Treating Ischemic Stroke
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AISCBF2025
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Acute Ischemic Stroke AIS
MeSH Terms: interventions — Galantamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- galantamine group (Experimental): Standard treatment for acute ischemic stroke and galantamine
  Interventions: Drug: Galantamine; Drug: Standard treatment for acute ischemic stroke
- Control group (Sham Comparator): Standard treatment for acute ischemic stroke
  Interventions: Drug: Standard treatment for acute ischemic stroke

INTERVENTIONS:
Drug: Galantamine — Start within 24 hours of hospitalization, administer 5.0 mg of galantamine via intramuscular injection once daily, and continue the treatment for 10 days.
  Other Names: Galantamine from Lycoris aurea extract
  Arms: galantamine group
Drug: Standard treatment for acute ischemic stroke — Standard treatment for acute ischemic stroke
  Other Names: Routine Western medical treatment according to guidelines

SUMMARY:
Although mechanical thrombectomy or thrombolytic therapy for large vessels can achieve a revascularization rate (TICI ≥2b) of over 90%, 30-50% of patients still exhibit poor functional outcomes. This phenomenon of "ineffective reperfusion" suggests that microcirculatory dysfunction plays a decisive role in post-stroke neural injury. Therefore, it is necessary to combine brain protection strategies with microcirculatory reperfusion therapy to improve the functional prognosis of stroke patients.Increasing cerebral blood flow (CBF) and neurovascular unit (NVU)-based cerebral protection are current hotspots in the emergency treatment of stroke.

Galantamine, extracted from Lycoris aurea (a traditional Chinese medicinal herb), is an acetylcholinesterase inhibitor (AChEI) that has been widely recognized for improving cerebral blood flow and modulating inflammatory responses in ischemic stroke (IS).

Therefore, the applicant will conduct an internationally compliant, randomized controlled clinical study with routine treatment to evaluate the efficacy of galantamine in the treatment of acute cerebral infarction. This project will conduct a comprehensive assessment of the drug's efficacy from multiple aspects, including improvements in stroke-related outcomes, Traditional Chinese Medicine (TCM) syndrome manifestations, cognitive function, cerebral blood flow, and inflammatory factors.

ELIGIBILITY:
Inclusion Criteria:

* Aged > 18 years and < 85 years, regardless of gender
* Meeting the diagnostic criteria for ischemic stroke in Western medicine
* Meeting the diagnostic criteria for stroke (Zhongfeng) in Traditional Chinese Medicine (TCM)
* Diagnosis of acute ischemic stroke within 72h of symptom onset
* A score of 4-25 points on the National Institute of Health Stroke Scale (NIHSS)
* First onset of the disease, or no severe sequelae related to previous onset
* The patient and their legal guardian voluntarily sign the informed consent form for the study

Exclusion Criteria:

* Confirmed by cranial imaging examination to have diseases causing similar symptoms such as brain tumors, encephalitis, and brain abscesses; or confirmed to have hemorrhagic cerebral infarction,epidural hematoma,intracranial hematoma, intraventricular hemorrhage, subarachnoid hemorrhage, etc.
* Patients with severe abnormalities of liver and kidney function (liver function: alanine aminotransferase [ALT] >2 times the upper limit of normal [ULN]; renal function: creatinine [Cr]>1.5 times the upper limit of normal [ULN])
* Elderly patients with physical weakness or patients complicated with infection
* Patients with a history of mental illness or dementia
* Patients with other severe organ or systemic diseases, accompanied by malignant tumors in any organ or system, or undergoing anti-tumor treatment, with an expected survival time of < 6 months
* A significant history of drug or alcohol abuse
* Women who test positive for blood human chorionic gonadotropin (HCG) (i.e., HCG ≥ 5 mIU/mL) during pregnancy screening, plan to become pregnant during the trial, or are breastfeeding
* Patients who are currently participating in other clinical trials or have participated in other clinical trials within the past 1 month
* Patients who are currently using other cholinesterase inhibitor drugs or have used other cholinesterase inhibitor drugs within the past 3 months
* Patients with epilepsy, hyperkinesis, mechanical intestinal obstruction, bronchial asthma, angina pectoris, bradycardia, or glaucoma
* Patients with contraindications to brain magnetic resonance imaging (MRI) examination, such as patients with implanted cardiac pacemakers, patients with implanted artificial joints or orthopedic plates, patients with claustrophobia, etc

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2028-09-14 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
The change in NIHSS score | Randomization Day,Day 10 (±2 days),Day 30 (±4 days) and Day 90 (±7 days)
  Scores on the National Institutes of Health Stroke Scale (NIHSS) range from 0 to 42, with higher scores indicating more severe neurologic deficits

SECONDARY OUTCOMES:
Scores assessed by Fugl-Meyer motor assessment (FMA) | Randomization Day,Day 10 (±2 days),Day 30 (±4 days) and Day 90 (±7 days)
  Scores on the Fugl-Meyer motor assessment (FMA) range from 0 to 100,with lower scores indicating more severe the motor dysfunction
Cerebral Blood Flow | Randomization Day,Day 30 (±4 days)
  The cerebral blood flow is evaluated by MRI
Fractional anisotropy (FA) values | Randomization Day,Day 30 (±4 days)
  The fractional anisotropy (FA) values is evaluated by MRI
TNF-α | Randomization Day,Day 10 (±2 days)
  Laboratory parameters obtained through venous blood analysis
IL-6 | Randomization Day,Day 10 (±2 days)
  Laboratory parameters obtained through venous blood analysis
Modified Rankin Scale (mRS) score | Randomization Day,Day 10 (±2 days),Day 30 (±4 days) and Day 90 (±7 days)
  The mRs is an ordinal disability score of 7 categories (0=no symptoms to 5=severe disability, and 6=death)
Scores assessed by Mini-Mental State Examination (MMSE) | Randomization Day,Day 10 (±2 days),Day 30 (±4 days) and Day 90 (±7 days)
  The MMSE is a brief 30-point questionnaire test that is used to screen for cognitive impairment. A score greater than or equal to 25 points is effectively normal (intact). Below this, scores can indicate severe (≤9 points), moderate (10-20 points) or mild (21-24 points) cognitive impairment
Scores assessed by Montreal Cognitive Assessment (MoCA) | Randomization Day,Day 10 (±2 days),Day 30 (±4 days) and Day 90 (±7 days)
  MoCA scores range between 0 and 30. Higher scores indicate a better outcome, and a score of 26 or over is considered to be normal
Traditional Chinese Medicine (TCM) syndrome manifestations | Randomization Day,Day 10 (±2 days),Day 30 (±4 days) and Day 90 (±7 days)
  Under the guidance of Traditional Chinese Medicine (TCM) theory, evaluate the drug's effect on improving TCM syndrome manifestations (such as hemiplegia, deviated mouth and tongue, and speech impairment).
Barthel Index Score | Randomization Day,Day 10 (±2 days),Day 30 (±4 days) and Day 90 (±7 days)
  It is used to measure the ability of patients (especially those with stroke, geriatric diseases, or in the rehabilitation period) to independently complete daily activities such as eating, dressing, walking, and using the toilet. The scoring range is 0-100 points, with higher scores indicating stronger self-care ability in daily life.
EQ-5D Scale Score | Randomization Day,Day 10 (±2 days),Day 30 (±4 days) and Day 90 (±7 days)
  It is an internationally accepted assessment tool for "Health-Related Quality of Life (HRQoL)". Its core function is to quantitatively evaluate an individual's health status and quality of life through five dimensions: "mobility, self-care, usual activities, pain/discomfort, and anxiety/depression". It is widely used in clinical trials, health economics research, and chronic disease management (e.g., comprehensive evaluation of treatment effects in stroke patients).

CONTACTS AND LOCATIONS:
Overall Officials: Chunxiang Chen, Study Chair — Shanghai Yueyang Integrated Medicine Hospital
Locations (1):
- Shanghai Yueyang Integrated Medicine Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No